CLINICAL TRIAL: NCT03838939
Title: Impact of Association of Individual and Group Therapeutic Education Sessions on the Acquisition of Safety Skills by Patients With Chronic Inflammatory Rheumatism (CIR) Treated With Subcutaneous Biotherapy, Compared to Individual Therapeutic Education Sessions Alone
Brief Title: Biotherapies and Therapeutic Education in Chronic Inflammatory Rheumatism
Acronym: ERIBIO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: French Society of Rheumatology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: CHU-420; 2018-A00647-48 (Other: 2018-A00647-48)
Record Dates: First submitted 2019-01-22; First posted 2019-02-12 (Actual); Last update posted 2021-12-22 (Actual); Status verified 2021-12

CONDITIONS: Rheumatoid Arthritis; Spondyloarthritis
Keywords: chronic inflammatory rheumatism; biotherapies; therapeutic education; safety skills
MeSH Terms: conditions — Arthritis, Rheumatoid; Spondylarthritis

STUDY DESIGN:
Masking Description: no masking
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- interventional group (Experimental): M3 (group with 3 to 10 patients) Intensification Biotherapy Education Workshops : "Subcutaneous injection education" and "biotherapy management
  Interventions: Other: Therapeutic education
- Control group (Placebo Comparator): M3 (individual) Intensification Biotherapy Education: "Subcutaneous injection education" and "biotherapy management".
  Interventions: Other: Therapeutic education

INTERVENTIONS:
Other: Therapeutic education — Individual and group therapeutic education sessions will consist of :
  * acquisition by patient of self-care skills such as performing subcutaneous injection,
  * acquisition by patient of safety skills such as identifying symptoms that should lead to consult general practitioner, and stop treatment ...

SUMMARY:
The hypothesis is that group interaction associated with individual interviews intensify the acquisition of safety skills compared to individual interviews alone in patients with CIR treated by subcutaneous biotherapies.

DETAILED DESCRIPTION:
Selection and inclusion of patients will be done by principal investigator of Rheumatology Department. After verification of inclusion and non-inclusion criteria by principal investigator and signature of consent, patients will be randomized by 1: 1 randomization (centralized randomization by statistician into 2 groups at M0) :

1. Experimental group (individual and group therapeutic education )

   * M0 (individual) Educational diagnosis and biotherapy education: "subcutaneous injection education" and "biotherapy management".
   * M3 (group with 3 to 10 patients) Intensification Biotherapy Education: Workshops : "Subcutaneous injection education" and "biotherapy management".
   * M6 (individual presential or by phone) Assessment of security skills and questionnaires.
   * M12 (individual presential or by phone) Assessment of security skills and questionnaires.
2. Control group (individual therapeutic education alone ) :

   * M0 (individual) Educational diagnosis and biotherapy education: "subcutaneous injection education" and "biotherapy management".
   * M3 (individual) Intensification Biotherapy Education: "Subcutaneous injection education" and "biotherapy management".
   * M6 (individual présential or by phone) Assessment of security skills and questionnaires.
   * M12 (individual présential or by phone) Assessment of security skills and questionnaires. Group session proposed.

ELIGIBILITY:
Inclusion Criteria:

* Patient age > 18 years old with RA (ACR/EULAR criteria) or SA (ASAS criteria) initiating a first subcutaneous biotherapy.
* Patient able to complete a questionnaire
* Patient giving informed consent.
* Patient covered by social security

Exclusion Criteria:

* - Patient with disorder of higher mental function or psychiatric disorders.
* Patient previously treated by intravenous biotherapy.
* Protected populations: pregnant women, breastfeeding women, tutorship, trusteeship, deprived of liberty, safeguard of justice.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2019-01-21 (Actual); Primary Completion 2021-12-10 (Actual); Study Completion 2021-12-10 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Biosecure's score at 6 months after biological treatment initiation | at 6 months
  Biosecure questionnaire assesses safety skills regarding infections, vaccinations, and situations of daily life (travel, surgery, pregnancy,…). It's composed of 29 questions about knowledge and 7 scenarios. The response methods are: yes / no / I don't know, with 55 items (score from 0 to 100 points), developed by Therapeutic Education Section of French Society of Rheumatology.

SECONDARY OUTCOMES:
Change from Baseline Biosecure's score at 6 months after biological treatment initiation | at 6 months
  Biosecure questionnaire assesses safety skills regarding infections, vaccinations, and situations of daily life (travel, surgery, pregnancy,…). It's composed of 29 questions about knowledge and 7 scenarios. The response methods are: yes / no / I don't know, with 55 items (score from 0 to 100 points), developed by Therapeutic Education Section French Society of Rheumatology.
Number of hospitalizations for infection during the year, collected from patient (tracking book) and in medical file, at the follow-up at M12 | at 12 months
  patient tracking book includes type of infection, stop biotherapy, consultation with attending physician, taking antibiotics, hospitalization and validation by treating physician
Number of biotherapy stops and number of visits to physician for infection, collected from patient at M6 and M12 (tracking book) | at 6 months and 12 months
  patient tracking book includes type of infection, stop biotherapy, consultation with attending physician, taking antibiotics, hospitalization and validation by treating physician
Type of infections occurring, collected from patient at M6 and M12 (tracking book ) | at 6 months and 12 months
  patient tracking book includes type of infection, stop biotherapy, consultation with attending physician, taking antibiotics, hospitalization and validation by treating physician
Coping evaluated by analogical visual scale at M6 and M12 | at 6 months and 12 months
  RAID questionnaire is calculated according to 7 numerical rating scales: pain, functional ability, fatigue, sleep, emotional well-being, physical well-being, and disease management. Each scale is evaluated by a number between 0 and 10. A final RAID score with high values characterize a disturbing state of the patient
Psychological well-being evaluated by Analogical visual scale at M6 and M12 by RAID questionnaire. | at 6 months and 12 months
  RAID questionnaire is calculated according to 7 numerical rating scales: pain, functional ability, fatigue, sleep, emotional well-being, physical well-being, and disease management. Each scale is evaluated by a number between 0 and 10. A final RAID score with high values characterize a disturbing state of the patient.
Fear about treatment evaluated by FAIR questionnaire at M6 and M12. | at 6 months and 12 months
  FAIR questionnaire (Fear Assessment in Inflammatory Rheumatic diseases) evaluate the levels of fear (side effects of treatment, disease progress,…) and psychological distress in patients, it be included in clinical trial protocols to measure the impact of specific interventions on psychological distress
Patient satisfaction evaluated with Patient satisfaction questionnaire | at 12 month
  Patient satisfaction questionnaire items are: overall satisfaction of education sessions, quality of content in line with expectations, teaching methods and tools used, course flow, quality of the exchange

CONTACTS AND LOCATIONS:
Overall Officials: Françoise FAYET, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- Chu Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Background] Gossec L, Fautrel B, Flipon E, Lecoq d'Andre F, Marguerie L, Nataf H, Pallot Prades B, Piperno M, Poilverd RM, Rat AC, Sadji F, Sordet C, Thevenot C, Beauvais C. Safety of biologics: elaboration and validation of a questionnaire assessing patients' self-care safety skills: the BioSecure questionnaire. An initiative of the French Rheumatology Society Therapeutic Education section. Joint Bone Spine. 2013 Oct;80(5):471-6. doi: 10.1016/j.jbspin.2012.11.009. Epub 2013 Aug 20. PMID 23972274
- [Background] Gronning K, Rannestad T, Skomsvoll JF, Rygg LO, Steinsbekk A. Long-term effects of a nurse-led group and individual patient education programme for patients with chronic inflammatory polyarthritis - a randomised controlled trial. J Clin Nurs. 2014 Apr;23(7-8):1005-17. doi: 10.1111/jocn.12353. Epub 2013 Jul 22. PMID 23875718
- [Background] Homer D, Nightingale P, Jobanputra P. Providing patients with information about disease-modifying anti-rheumatic drugs: Individually or in groups? A pilot randomized controlled trial comparing adherence and satisfaction. Musculoskeletal Care. 2009 Jun;7(2):78-92. doi: 10.1002/msc.141. PMID 18792423
- [Background] Koev DJ, Tankova TI, Kozlovski PG. Effect of structured group education on glycemic control and hypoglycemia in insulin-treated patients. Diabetes Care. 2003 Jan;26(1):251. doi: 10.2337/diacare.26.1.251. No abstract available. PMID 12502698
- [Derived] Fayet F, Beauvais C, Pereira B, Beranger M, Rodere M, Pallot-Prades B, Peyrard P, Pouplin S, Grandjean M, Chu Miow Lin D, Ardizzone M, Cherillat MS, Tournadre A, Fan A, Soubrier M. Comparison of group versus individual patient education for promoting safety skills of patients with autoimmune rheumatic diseases treated with biologics: a multicentre randomised controlled trial. Clin Rheumatol. 2025 Jan;44(1):487-494. doi: 10.1007/s10067-024-07218-6. Epub 2024 Nov 5. PMID 39499437